CLINICAL TRIAL: NCT07014982
Title: Remote Assessment of Digital Neurologic Testing (RADiaNT)
Brief Title: Remote Assessment of Digital Neurologic Testing
Acronym: RADiaNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David T. Jones, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-013687
Record Dates: First submitted 2025-05-15; First posted 2025-06-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Neurology
Keywords: Neurology

STUDY DESIGN:
Intervention Model Description: This study will have two cohorts; one intervention cohort and one control cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Meditation (Experimental): This cohort will be practicing guided meditation for 5 days/week, five minutes a day for 6 weeks. Then there will be a period of testing followed by another 6 week period of practicing guided meditation.
  Interventions: Behavioral: Guided Meditation
- Standard of Care (No Intervention): This cohort will be asked to complete neurologic testing at baseline, interim, and conclusion periods while conducting NO guided meditation throughout the duration of the study.

INTERVENTIONS:
Behavioral: Guided Meditation — Participants who complete guided meditation will be asked to meditate for 5 minutes a day, five times a week for two 6-week periods.
  Arms: Guided Meditation

SUMMARY:
The RADiaNT study investigates whether guided meditation, using the Muse™ headband and biofeedback app, can improve sleep, mood, and cognitive performance, aiming to assess its impact on mental and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Cognition unimpaired or mild cognitive impairment
* Fluent in English
* United States resident
* Able to tolerate wearing Muse headband
* basic competence in using electronic devices (Smartphone or tablet) to engage with the Muse application and complete digital surveys and assessments

Exclusion Criteria:

* Neurological and Brain Disorders
* Not Fluent in English
* Not a US Resident
* Unable to tolerate wearing Muse Headband

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Duration in slow wave sleep | 17 weeks
  Total duration of sleep time spent in slow wave sleep (delta), reported in minutes
Proportion in slow wave sleep | 17 weeks
  Proportion is the percentage of sleep time spent in slow wave sleep (delta)
Perceived Stress Scale | 17 weeks
  Investigators will ask patients to answer the PSS questionnaire at the beginning, interim, and end of the study to see if there were any improvements in sleep quality over the intervention periods. This questionnaire is on a scale that scores 0-40, with the higher the score being a higher level of stress.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | 17 weeks
  The Patient Health Questionnaire 9-item (PHQ-9) scale used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.
General Anxiety Disorder 7-item (GAD-7) | 17 weeks
  The General Anxiety Disorder 7-item (GAD 7) scale to assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety.
Cognitive Performance | 17 weeks
  Investigators will test patients' cognitive performance at the beginning, interim, and conclusion of the study using Mayo Speech Test.
Cognitive Performance | 17 weeks
  Investigators will test patients' cognitive performance at the beginning, interim, and conclusion of the study using Mayo Test Drive.

CONTACTS AND LOCATIONS:
Overall Officials: David Jones, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No